CLINICAL TRIAL: NCT05157191
Title: A Prospective Observational Study to Evaluate the Safety of COVID-19 Vaccination in Children and Adolescents
Brief Title: Safety of Pediatric COVID-19 Vaccination
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Kaiser Permanente (Other); Columbia University (Other); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00110056
Record Dates: First submitted 2021-12-10; First posted 2021-12-14 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Pain; Injection Site Reaction; Adverse Drug Event
Keywords: COVID-19 vaccine; fever following vaccination; pain following vaccination
MeSH Terms: conditions — Pain; Injection Site Reaction; Drug-Related Side Effects and Adverse Reactions | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- mRNA COVID-19 vaccine: Children and adolescents (ages ≥ 5 to < 16) who receive mRNA COVID-19 vaccine per standard of care
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational

SUMMARY:
This is a prospective, observational study. During the study, children and adolescents (ages ≥ 5 to < 16) will be followed post administration of mRNA COVID-19 vaccines.

Injection site (local), systemic reaction, and unsolicited adverse event data will be assessed on vaccination day and during the 7 days following each vaccination using either identical web-based or paper diaries, depending on study participant preference.

At Duke University, Cincinnati's Children Hospital, and Kaiser Permanente Northern California, serum samples will be collected for optional assessment of antibody titers to COVID-19. Each participant who opts in will have baseline (within 3 days of vaccination) serologies obtained and immunogenicity assessment at 28 (+7) days after each dose.

All participants will be followed for 180 days after dose 2 for serious adverse events and adverse events of special interest.

ELIGIBILITY:
Inclusion Criteria:

1. Children ≥ 5 years to < 16 years of age
2. Receiving first dose or a booster dose of a U.S authorized or approved and recommended COVID-19 vaccine per standard of care
3. Parent/legal authorized representative (LAR) willing to provide written informed consent per local IRB requirements
4. Participant willing to provide assent per local IRB requirements
5. Intention of being available for entire study period and complete all relevant study procedures, including follow-up phone calls
6. English or Spanish literate.

Exclusion Criteria:

1. Current or planned participation in any clinical trial with an investigational product during the study period.*

   * Per protocol, co-enrollment in observational or behavioral intervention studies are permitted at any time. An investigational product or behavioral intervention permitted at any time. An investigational product may be permitted for therapy of an illness condition that occurs during the study period (e.g., COVID-19 illness)
2. Any condition, which, in the opinion of the investigators, may pose a health risk to the subject or interfere with the evaluation of the study objectives.
3. Anyone who is a relative of any research study personnel or is an employee supervised by study staff.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 320 healthy male or female ≥ 5 years to < 16 years of age
Sampling Method: Non-Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
Number of participants with defined local or systemic reactogenicity events after each dose of COVID-19 vaccine | Up to 7 days post-vaccination
  Tables summarizing each solicited local and systemic reactogenicity event by maximum classification (none, mild, moderate, and severe), as well as by moderate or severe
Number of participants with at least one severe (Grade 3) solicited local or systemic reactogenicity event after each dose of COVID-19 vaccine | Up to 7 days post-vaccination
  Tables summarizing each severe (Grade 3) solicited local and systemic reactogenicity event
Number of participants with at least one moderate-to-severe (Grade 2-3) solicited local or systemic reactogenicity event after each dose of COVID-19 vaccine | Up to 7 days post-vaccination
  Tables summarizing each moderate-to-severe (Grade 2-3) solicited local and systemic reactogenicity event
Number of participants with an unsolicited adverse events after each dose of COVID-19 vaccine | Up to 7 days post-vaccination
  The number and percent and descriptions of unsolicited adverse events observed
Number of participants with an adverse event of special interest | Up to 29 days post-vaccination
  The number and percent of individuals with an adverse event of special interest after dose 2 of COVID-19 vaccine
The number and percent of participants with at least one serious adverse event after dose 2 of COVID-19 vaccine | Up to 29 days post-vaccination
  The number and percent of serious adverse events observed and description of each event

SECONDARY OUTCOMES:
Number of participants with defined local or systemic reactogenicity events after receiving other routinely recommended vaccines with each dose of COVID-19 vaccine | Up to 7 days post-vaccination
  Tables summarizing each solicited local and systemic reactogenicity event by maximum classification (none, mild, moderate, and severe), as well as by moderate or severe
Number of participants with defined local or systemic reactogenicity events after receiving each dose of COVID-19 vaccine without other vaccines | Up to 7 days post-vaccination
  Tables summarizing each solicited local and systemic reactogenicity event by maximum classification (none, mild, moderate, and severe), as well as by moderate or severe
Number of participants with at least one severe (Grade 3) solicited local or systemic reactogenicity event after other routinely recommended vaccines with each dose of COVID-19 vaccine | Up to 7 days post-vaccination
  Tables summarizing each moderate to severe (Grade 2-3) solicited local and systemic reactogenicity event
Number of participants with at least one severe (Grade 3) solicited local or systemic reactogenicity event after receiving COVID-19 vaccine without receiving other vaccines | Up to 7 days post-vaccination
  Tables summarizing each severe (Grade 3) solicited local and systemic reactogenicity event
Number of participants with at least one moderate-to-severe (Grade 2-3) solicited local or systemic reactogenicity event after receiving other routinely recommended vaccines with each dose of COVID-19 vaccine | Up to 7 days post-vaccination
  Tables summarizing each moderate-to-severe (Grade 2-3) solicited local and systemic reactogenicity event
Number of participants with at least one moderate-to-severe (Grade 2-3) solicited local or systemic reactogenicity event after receiving COVID-19 vaccine without receiving other vaccines | Up to 7 days post-vaccination
  Tables summarizing each moderate-to-severe (Grade 2-3) solicited local and systemic reactogenicity event
Number of participants with an unsolicited adverse events after receiving other routinely recommended vaccines with each dose of COVID-19 vaccine | Up to 7 days post-vaccination
  The number and percent and descriptions of unsolicited adverse events observed
Number of participants with an unsolicited adverse events after receiving other routinely recommended vaccines with each dose of COVID-19 vaccine without receiving other vaccines | Up to 7 days post-vaccination
  The number and percent and descriptions of unsolicited adverse events observed
Number of participants with an adverse event of special interest who received other routinely recommended vaccines with each dose of COVID-19 vaccine | Up to 29 days post-vaccination
  The number and percent of individuals who had at least one adverse event of special interest
Number of participants with an adverse event of special interest who received other routinely recommended vaccines with each dose of COVID-19 vaccine without receiving other vaccines | Up to 29 days post-vaccination
  The number and percent of individuals who had at least one adverse event of special interest
The number and percent of participants with at least one serious adverse event who received other routinely recommended vaccines after dose 2 of COVID-19 vaccine | Up to 29 days post-vaccination
  The number and percent of serious adverse events observed and description of each event
The number and percent of participants with at least one serious adverse event who received other routinely recommended vaccines after dose 2 of COVID-19 vaccine without receiving other vaccines | Up to 29 days post-vaccination
  The number and percent of serious adverse events observed and description of each event

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Smith, MD, Principal Investigator — Duke University
Locations (5):
- United States (5):
  - Kaiser Permanente Northern California, Oakland, California
  - Centers for Disease Control and Prevention, Atlanta, Georgia
  - Columbia University, New York, New York
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-03): https://cdn.clinicaltrials.gov/large-docs/91/NCT05157191/Prot_SAP_001.pdf